CLINICAL TRIAL: NCT04204304
Title: The Relationship Between Serum 25 Hydroxy Vitamin D Levels and Musculoskeletal Adverse Effects in Patients With Acne Vulgaris Using Isotretinoin: A Cross-sectional Controlled Study
Brief Title: Relationship Between Serum Vitamin D Levels and Musculoskeletal Adverse Effects in Patients Using Isotretinoin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cevriye Mülkoğlu, Director, clinical research, Ankara Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AnkaraTRH
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Musculoskeletal Disease Other; Isotretinoin Adverse Reaction; Vitamin D Deficiency
Keywords: D014807; D02.455.326.271.665.202.495.325; C17.800.030.150
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isotretinoin-induced adverse effect group (Experimental): Patients receiving isotretinoin with dose of 0.5-1 mg/kg/day and had musculoskeletal adverse effects
  Interventions: Drug: Isotretinoin
- Control group (Active Comparator): Pateients receiving isotretinoin with dose of 0.5-1 mg/kg/day had no musculoskeletal adverse effects
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — ISO
  Other Names: Isotretinoin capsules

SUMMARY:
Isotretinoin (ISO) has been used in the treatment of patients with severe acne vulgaris (AV) that is resistant to standard therapy with systemic antibiotics and topical agents, over the last few decades. There are various side effects of ISO in the skeletal system.

This study investigate the relationship between ISO-induced musculoskeletal adverse effects and serum 25 hydroxy (OH) vitamin D levels in patients with acne vulgaris.

DETAILED DESCRIPTION:
The rheumatic side effects are the most common one which are musculoskeletal pains and arthralgia, seen over of the 16% patients receiving ISO. Mild, transient myalgias and arthralgias are very common and do not require cessation of the drug. The other musculoskeletal side effects of ISO are calcification of tendon and ligaments, hyperostosis of the spine (DISH syndrome), elevated creatine phosphokinase and cramps. There are many case reports related with ISO-induced sacroiliitis in the literature, mostly recent years.

The association between ISO and vitamin D levels has been evaluated with several studies in the literature17,18,19. However, the relationship between ISO-induced musculoskeletal side effects in AV patients and serum vitamin D levels has not been investigated until now. To the best our knowledge, this is the first study to evaluate the relationship between the serum vitamin D levels and the musculoskeletal side effects related with ISO in AV patients.

In this study, 87 patients receiving ISO for AV and had ISO-induced musculoskeletal side effects, were enrolled as adverse effect (AE) group. The control (C) group was consisted of age- and sex-matched 90 consecutive patients using ISO but had no musculoskeletal symptoms.

The participants was assessed in aspect of musculoskeletal symptoms such as arthralgia, low back pain, calsification of tendon and ligaments, polyneuropathy, hyperostoses of the spine (DISH syndrome), myalgia, cramps and sacroiliitis. It was queried that whether myalgia, arthralgia, low back pain or sacroiliitis has occurred after ISO treatment. Serum 25 (OH) vitamin D levels were measured in all participants. According to these results, patients in AE group were divided into three subgroups in aspect of the serum vitamin D levels. Patients with serum 25 (OH) vitamin D level is lower than 10 ng/ml, was recruited as Group I, between 10-20 ng/ml, as Group II, higher than 20 ng/ml as Group III.

ELIGIBILITY:
Inclusion Criteria:

* ISO at a dose of 0.5-1 mg/kg/day for at least 3 months,
* not to use vitamin D and/or calcium supplements for the last three months
* to be older than 18 years.

Exclusion Criteria:

* Patients who had renal, gastroenteritis, skeletal, psychiatric, hematological, endocrine disorders related with thyroid and bone metabolism
* Patients receiving drugs such as diuretics, multivitamins, anticonvulsants, glucocorticoids, erythromycin, estrogen compound pills, alcohol, vitamin D and/or calcium preparats in the last three months,
* Malignancy,
* Chronic liver and kidney failure,
* History of psoralen and ultraviolet A (PUVA)
* Women waiting pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal adverse effects in isotretinoin receiving patients | 2 days
  Locomotor system examination of the participants will perform by the same clinician.The participants were assessed in aspect of musculoskeletal symptoms such as arthralgia, low back pain, calcification of tendon and ligaments, polyneuropathy, hyperostoses of the spine (DISH syndrome), myalgia, cramps and sacroiliitis
Serum 25 hydroxy vitamin D level | 7 days
  serum vitamin d levels will measure in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Cevriye Mülkoğlu, Principal Investigator — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No